CLINICAL TRIAL: NCT01163877
Title: Iron Absorption and Utilization in Adolescents Infected With Malaria Parasites, Hookworms or Schistosoma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EK-2009-N-19
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Malaria, Falciparum; Hookworm Infections; Schistosoma Haematobium
Keywords: iron absorption; iron utilization; malaria; helminth; Ivory Coast; Acute symptomatic uncomplicated falciparum malaria; Asymptomatic falciparum malaria; Moderate to heavy hookworm infection; Heavy Schistosoma haematobium infection
MeSH Terms: conditions — Malaria, Falciparum; Hookworm Infections; Schistosomiasis haematobia; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Symptomatic malaria infection (Other)
  Interventions: Dietary Supplement: Fe-57 orally, Fe-58 intravenously
- Asymptomatic malaria infection (Other)
  Interventions: Dietary Supplement: Fe-57 orally, Fe-58 intravenously
- Hookworm infection (Other)
  Interventions: Dietary Supplement: Fe-57 orally, Fe-58 intravenously
- Schistosoma haematobium infection (Other)
  Interventions: Dietary Supplement: Fe-57 orally, Fe-58 intravenously

INTERVENTIONS:
Dietary Supplement: Fe-57 orally, Fe-58 intravenously — Subjects will receive a test drink containing 3 mg Fe-57 in the form of labelled FeSO4 followed by 1 ml of an aqueous solution containing 50 μg Fe-58 as iron citrate.

SUMMARY:
The aim of this study is to investigate the change in iron metabolism in relation to malaria and helminth infections using a stable isotope technique.

DETAILED DESCRIPTION:
The aim of the study is to determine how iron metabolism in subjects with infectious diseases (malaria, hookworm or S. haematobium) differs while infected and after treatment, i.e. the same individuals will be restudied while free of infection.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12 to 16 years
* Body weight > 30 kg
* no chronic medical illnesses
* no intake of vitamin/mineral supplements 2 weeks before the study and until the last blood drawing
* For each of the 4 arms the respective disease needs to be present (symptomatic malaria, asymptomatic malaria, hookworm infection, S. haematobium infection) without any other concurrent infection

Exclusion Criteria:

-

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2010-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Isotope absorption into blood stream | Day 15
Isotope absorption into blood stream | Day 43

SECONDARY OUTCOMES:
Isotope incorporation into erythrocytes | Day 15
Biochemical parameters of iron status and infection | Day 1
Biochemical parameters of iron status and infection | Day 15
Biochemical parameters of iron status and infection | Day 29
Biochemical parameters of iron status and infection | Day 43
Isotope incorporation into erythrocytes | Day 43

CONTACTS AND LOCATIONS:
Overall Officials: Rita Wegmüller, Dr., Principal Investigator — Swiss Federal Institute of Technology (ETH) Zurich
Locations (1):
- Taabo Cité Hospital, Taabo, Côte d’Ivoire

REFERENCES:
- [Background] Rohner F, Zimmermann MB, Amon RJ, Vounatsou P, Tschannen AB, N'goran EK, Nindjin C, Cacou MC, Te-Bonle MD, Aka H, Sess DE, Utzinger J, Hurrell RF. In a randomized controlled trial of iron fortification, anthelmintic treatment, and intermittent preventive treatment of malaria for anemia control in Ivorian children, only anthelmintic treatment shows modest benefit. J Nutr. 2010 Mar;140(3):635-41. doi: 10.3945/jn.109.114256. Epub 2010 Jan 27. PMID 20107144
- [Background] Wegmuller R, Camara F, Zimmermann MB, Adou P, Hurrell RF. Salt dual-fortified with iodine and micronized ground ferric pyrophosphate affects iron status but not hemoglobin in children in Cote d'Ivoire. J Nutr. 2006 Jul;136(7):1814-20. doi: 10.1093/jn/136.7.1814. PMID 16772442
- [Background] Kastenmayer P, Davidsson L, Galan P, Cherouvrier F, Hercberg S, Hurrell RF. A double stable isotope technique for measuring iron absorption in infants. Br J Nutr. 1994 Mar;71(3):411-24. doi: 10.1079/bjn19940148. PMID 8172870
- [Background] Walczyk T, Davidsson L, Zavaleta N, Hurrell RF. Stable isotope labels as a tool to determine the iron absorption by Peruvian school children from a breakfast meal. Fresenius Journal of Analytical Chemistry 359: 445-449, 1997.
- [Derived] Glinz D, Hurrell RF, Righetti AA, Zeder C, Adiossan LG, Tjalsma H, Utzinger J, Zimmermann MB, N'Goran EK, Wegmuller R. In Ivorian school-age children, infection with hookworm does not reduce dietary iron absorption or systemic iron utilization, whereas afebrile Plasmodium falciparum infection reduces iron absorption by half. Am J Clin Nutr. 2015 Mar;101(3):462-70. doi: 10.3945/ajcn.114.090175. Epub 2015 Feb 4. PMID 25733630